CLINICAL TRIAL: NCT01501292
Title: Changes in the Distribution of Mitochondria During Oocyte Maturation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0095-11-HYMC
Record Dates: First submitted 2011-12-13; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Staining and Labeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Immature oocytes (GV, M-I)
  Interventions: Other: Fixation and staining; Other: Observation by laser microscopy
- Mature oocytes (M-II)
  Interventions: Other: Fixation and staining; Other: Observation by laser microscopy

INTERVENTIONS:
Other: Fixation and staining — Fixation and staining by MitiTracker Green FM
Other: Observation by laser microscopy — Observation with Laser scanning confocal microscopy

SUMMARY:
Cytoplasmatic maturation is an important event in the general maturation of of the oocyte. Mitochondria is one of the major organelles involved in the process of cytoplasmatic maturation. The aim of this study is to investigate the presence and distribution of the mitochondria in the cytoplasma of immature oocytes that are retrieved in the routine in-vitro maturation cycle with intracytoplasmatic sperm injection (ICSI). These oocytes will not undergo ICSI because of their immaturity. Usually, they are discarded. In addition to these immature oocytes the investigators shall also investigate the mitochondria in mature oocytes that underwent ICSI but did not become fertilized and are discarded.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients needing IVF treatment

Exclusion Criteria:

* Patients not requiring the ICSI procedure

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing routine in-vitro fertilization with ICSI
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
The patterns of mitochondrial distribution within the cytoplasma of oocytes during nuclear maturation | Three months
  Identification the different patterns of mitochondrial distribution in correlation with the 3 stages nuclear maturation in human oocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel